CLINICAL TRIAL: NCT06740461
Title: The Correlation Between Ambulatory Blood Pressure Control and Aortic Stiffness Index Assessed by CMR After Aortic Coarctation Stenting in Adults
Brief Title: Aortic Stiffness by CMR in Aortic Coarctation
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shady Elia Ramzy, Resident doctor, Assiut University
Other Study IDs: Aortic stiffness by CMR in CoA
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Aortic Coarctation
Keywords: Aortic coarctation; Aortic stiffness; CMR; Ambulatory blood pressure
MeSH Terms: conditions — Aortic Coarctation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aortic coarctation patient

SUMMARY:
This study investigates the correlation between medium-term systemic blood pressure control and aortic stiffness index in adults following coarctation stenting, using cardiac magnetic resonance (CMR) imaging.

DETAILED DESCRIPTION:
Coarctation of the aorta (COA) is a common form of congenital heart disease with an incidence of 1 in 3000-4000 live births, characterized by the narrowing of the aorta, which leads to significant hemodynamic changes, including increased afterload, hypertension, and ultimately, adverse cardiovascular outcomes.

Despite successful surgical or interventional treatment to correct the anatomical defect, patients with coarctation of the aorta often continue to experience elevated systemic blood pressure and increased aortic stiffness, which are important predictors of long-term cardiovascular morbidity and mortality.

Stenting has emerged as a preferred interventional strategy for treating aortic coarctation in adults due to its less invasive nature and immediate efficacy in relieving aortic obstruction.

However, the medium-term impact of stenting on aortic stiffness remains underexplored. Understanding these changes is crucial for optimizing long-term management strategies and improving patient outcomes.

Cardiac magnetic resonance (CMR) imaging offers a non-invasive and highly accurate method for assessing aortic stiffness, providing detailed insights into the structural and functional properties of the aorta. The aortic stiffness index, derived from CMR measurements, serves as a valuable biomarker for vascular health and has been linked to systemic blood pressure levels.

This study aims to investigate the correlation between medium-term systemic blood pressure control and aortic stiffness index in adults following coarctation stenting.

By assessing patients pre- and post-stenting using CMR, we seek to determine whether improvements in aortic stiffness correspond with better blood pressure management over time. Our findings could provide valuable insights into the benefits of stenting beyond immediate hemodynamic relief, highlighting its role in the long-term cardiovascular health of patients with aortic coarctation.

ELIGIBILITY:
Patient criteria Inclusion criteria All patients with native or recurrent aortic coarctation between the age of 14 years and older.

Transcatheter systolic gradient ≥ 20 mm Hg, body weight ≥ 20 kg, and normal LV ejection fraction (EF).

Exclusion criteria Patients with obstructive lesion of LVOT or aortic valve dysfunction greater than moderate (requiring surgical intervention).

Irregular cardiac rhythm. Patients with other causes of secondary hypertension. Contraindications to CMR: Any contraindications to undergoing CMR, such as implanted metallic devices incompatible with MRI, severe claustrophobia.

Unicuspid aortic valve Associated complex congenital heart defects (aside from simple septal defects and patent ductus arteriosus) Genetic syndromes Connective tissue disorder History of surgery involving the aortic root or ascending aorta.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient with aortic coarctation undergoing transcatheter aortic stenting
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Correlation Between Systemic Blood Pressure and Aortic Stiffness Index | 1 year
  Evaluate the correlation between changes in systemic blood pressure and changes in the aortic stiffness index.
Change in Systemic Blood Pressure | 1 year
  Measure the change in systemic blood pressure (both systolic and diastolic) by ambulatory blood pressure for 24 hours.
Change in Aortic Stiffness Index | 1 year
  Measure the change in aortic stiffness index (derived from CMR) from baseline to the medium-term follow-up period.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lane DA, Lip GY, Millane TA. Quality of life in adults with congenital heart disease. Heart. 2002 Jul;88(1):71-5. doi: 10.1136/heart.88.1.71. PMID 12067950
- [Background] Ringel RE, Vincent J, Jenkins KJ, Gauvreau K, Moses H, Lofgren K, Usmani K. Acute outcome of stent therapy for coarctation of the aorta: results of the coarctation of the aorta stent trial. Catheter Cardiovasc Interv. 2013 Oct 1;82(4):503-10. doi: 10.1002/ccd.24949. Epub 2013 May 15. PMID 23592408
- [Background] Vonder Muhll IF, Sehgal T, Paterson DI. The Adult With Repaired Coarctation: Need for Lifelong Surveillance. Can J Cardiol. 2016 Aug;32(8):1038.e11-5. doi: 10.1016/j.cjca.2015.12.036. Epub 2016 Jan 21. PMID 27084076
- [Background] Grech V. Diagnostic and surgical trends, and epidemiology of coarctation of the aorta in a population-based study. Int J Cardiol. 1999 Feb 28;68(2):197-202. doi: 10.1016/s0167-5273(98)00352-0. PMID 10189008